

## PIETRO ARAÚJO DOS SANTOS

# NINTENDO WII AND EXERCISES AT REHABILITATION OF INDIVIDUALS WITH PARKINSON'S DISEASE

### **INFORMED CONSENT FORM**

NCT03235284

Salvador

11/09/2019



All the measurement instruments used in this study are documented as valid and reliable in Brazil. The study was approved by the ethics committee of the Health Sciences Institute of UFBA (under registration number CAAE: 41572914.5.0000.5662), in which all the participants signed the informed consent form.

#### **INFORMED CONSENT FORM**

We are pleased to invite you to participate in the research project titled: COMPARISON BETWEEN THE EFFECTS OF A TRAINING BASED ON THE FNP METHOD AND VIRTUAL REHABILITATION IN THE TREATMENT OF PATIENTS WITH PARKINSON'S DISEASE, under the responsibility of the researcher: Ms. Nildo Ribeiro. We report that the main objective of this research is to evaluate the effects of exercises performed through the PNF method and virtual rehabilitation in the treatment of patients with Parkinson's disease and the impact on quality of life. His evaluation will be carried out at the Professor Francisco Magalhães Neto Ambulatory, located at Rua Augusto Viana, s / n, Canela, Canela University Campus of the HUPES Complex, CEP:

40110-060, Salvador, Bahia. Data will be collected between August 2015 and August 2017. Their participation consists in making an evaluation to verify their functional independence, encompassing their ability to perform daily activities and answer questionnaires about their limitations and quality of life.

#### Discomfort and Possible Risks associated with the research:

The possible discomfort is associated with the evaluation and treatment procedures that can generate fatigue and the risk corresponding to fall, however the place will be adapted with stairs and ramps with handrail and non-slip floor, in the possibility of minimizing such risk. You will be accompanied by trained professionals throughout the time of your participation, and you may discontinue the evaluation or treatment at any time when you feel tired or uncomfortable. In addition you should report any type of discomfort felt during the research.

#### RESEARCH BENEFITS:

To determine the effectiveness of the techniques, NPF, this being a physiotherapy technique that aims at neuroproprioceptive facilitation and Nintendo Wii, this being an electronic game, focusing on the rehabilitation of patients with PD, enabling health professionals to develop strategies and programs for prevention and / or rehabilitation for the entire population, bringing benefits to society.

#### Accompaniment and Assistance Form:

The risks in the execution of the project will be minimized, but if necessary, you will receive all the health and / or social assistance to the aggravations resulting from the research activities and in the case of an emergency the Mobile Emergency Service of the city of Savior. However, any questions may be addressed to the researcher Nildo Ribeiro, at work phone 71-32838123 or personal 71-8194-1458 and by e-mail: nildoribeiro67@gmail.com

#### **CLARIFICATIONS AND RIGHTS**

At any time you can obtain clarification on all the procedures used in the research and on the ways of disseminating the results. You will have the freedom and right to refuse your participation or withdraw your consent at any stage of the research, without prejudice to the usual care provided by

| the research | chers. I | f you hav | e questions about | your particip | ation in the | e research you should co | ntact the |
|---|---|---|---|---|---|---|---|
| responsib | le resea | rcher at: | Health Sciences | Institute at A | Av. Rector | Miguel Calmon s / n - | Vale do |
| Canela | 4th | floor, | Physiotherapy | college | (71- | 32838914/81941458) | emai |
| nildoribei | ro67@g | gmail.con | n | | | | |

Voluntary nature of the study / Freedom to withdraw

Your participation is voluntary and you have the right to refuse to participate for any reason and withdraw your consent at any stage of the research, without any penalty and without prejudice to your care.

#### Confidentiality and evaluation of records

Ms. Nildo Ribeiro

Your identity will be kept in full secrecy for an indefinite period, both by the executor and by the institution where it will be held. The results of the procedures performed in the research will be analyzed and allocated to tables, figures or graphs and disseminated in lectures, conferences, scientific journals or other forms of dissemination that allow the transfer of knowledge to society and national or international health regulatory authorities, in accordance with the rules / statutory laws of national or international protection.

You will also receive a report at the end of the survey informing you about your evaluation and the results of this evaluation

| Post-Information Consent |
|---|
| . bearer of Identity Card |
| No, bearer of Identity Card, for considering me duly |
| informed and clarified on the content of this term and the research to be developed, freely expressing |
| my consent for inclusion, as subject the research. All information provided by me and the results |
| obtained will be kept confidential and the latter will be used for dissemination in meetings and |
| scientific journals without my identification. I will be informed of all the results obtained, regardless |
| of whether I change my consent to participate in the research. I will not have any financial benefits |
| or rights on the possible results of the research. I have been informed that my registration number in |
| the survey is and I received a copy of this document that I signed. |
| Signature of Participant Volunteer Date |
| Signature of Latticipant Volunteer Date |

Date